## Informed Consent Form (Parent/Guardian)

in relation to the research project: "Developing Innovative PTSD Treatment for Children: Reconsolidation of Traumatic Memories Protocol<sup>TM</sup> for Children (RTM-C Protocol)"

| I, | | , have | read | and understood | d the Parent Memo | o reg | garding the al | bove- |
|---|---|---|---|---|---|---|---|---|
| mentio | ned research pr | oject conduct | ed by | the research te | eam from the Glob | al I | nstitute for M | [ental |
| Health | Innovations, | Networking | and | Development | (GlobalInMind), | in | partnership | with |
| Charita | ble Foundation | Voices of Ch | ildren | (Ukraine) and | Quresta, Inc. (USA | <b>A</b> ). | | |

I have been informed both orally and in writing about the nature, purpose, duration, procedures, potential risks, and benefits of participating in the project, and I have had the opportunity to ask questions. I understand that participation is voluntary, and I may withdraw my consent at any time without giving reasons. If withdrawn, my child will be offered another method and referred if needed.

## I have been informed that:

- My personal data and my child's data will be processed in accordance with the Law of Ukraine on the Protection of Personal Data.
- All data will be anonymized by an RTM specialist.
- No identifying data will be shared. I may access, correct, or delete data.

## Please indicate your consent below:

| Statement | Yes | No |
|---|---|---|
| I consent to participate in this research study, including completing questionnaires. | | |
| I agree my child to participate (incl. RTM-C Protocol sessions, questionnaires). | | |
| I agree that my anonymised data can be used for scientific publications. | | |
| I agree to the data I provide being archived and used in anonymized form for other | | |
| I voluntarily agree (for me and my child) to take part in the Lux4UA Project. | | |

| Parent/guardi | an name: | | |
|---|---|---|---|
| Email: | Phone: | | |
| Date, place: | | _ | |
| Signature: | | | |
| RTM Special | ist statement: | | |
| I explained th | ne purpose, procedures, ris | sks, and benefits, and answered question | ıs. |
| Name: | Date, place: | Signature: | |

Responsible researcher: Viktoria Horbunova

Emails: viktoriyka.gorbunova@gmail.com, institute@globalinmind.eu Phone: +38 093 131 63 22, +33 9 74 06 34 21

GlobalinMind: https://www.globalinmind.eu Voices of Children: https://voices.org.ua

Post Traumatic Training Institute: https://thertmprotocol.com